CLINICAL TRIAL: NCT00995410
Title: A 12-Month, Phase 3, Open-Label, Multi-Center Study to Evaluate the Long-Term Safety of PA32540 in Subjects Who Are at Risk for Developing Aspirin-Associated Gastric Ulcers
Brief Title: Study to Evaluate the Long-Term Safety of PA32540 in Subjects Who Are at Risk for Developing Aspirin-Associated Gastric Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA32540-303
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Aspirin-Associated Gastric Ulcers
Keywords: Subjects Who are at Risk for Developing Aspirin-ASA; Subject must have a pre-existing condition for which aspirin is already indicated; Gastric Ulcers
MeSH Terms: conditions — Stomach Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PA32540 tablet (Experimental): 325 mg enteric coated (EC) ASA and 40 mg omeprazole to be taken by mouth once daily
  Interventions: Drug: PA32540

INTERVENTIONS:
Drug: PA32540 — PA32540 tablets contain 325 mg enteric coated (EC) aspirin and 40 mg immediate-release omeprazole to be taken by mouth once daily
  Other Names: YOSPRALA

SUMMARY:
This study uses an open-label design and will be conducted in approximately 40 sites in the United States. Approximately 400 subjects will be enrolled in the study to ensure that approximately 300 subjects will have 6 months exposure to PA32540 and at least 100 subjects will have 12 months exposure to PA32540.

DETAILED DESCRIPTION:
PA32540 is proposed for the secondary prevention of cardio- and cerebrovascular events in patients at risk for developing aspirin-associated gastric ulcers. This study is designed to provide long-term safety data for PA32540 in order to gain regulatory approval to make PA32540 available for clinical use in this subject population.

ELIGIBILITY:
Inclusion criteria:

1. A. Male or non-pregnant, non-breastfeeding females who have been on daily aspirin 325 mg for at least three months and who are expected to use daily aspirin 325 mg for at least six months (Daily is defined as "at least 5 days per week"):

   AND, who are
   * 55 years of age and older; or
   * 18 - 54 years of age and have a history of a documented gastric or duodenal ulcer within the past five years.
2. A. Aspirin use should be for the secondary prevention of cardiovascular or cerebrovascular events as defined as follows:

   Have been diagnosed with or have had a history of
   * MI (myocardial infarction that has been confirmed or suspected)
   * Ischemic stroke
   * TIA (transient ischemic attack)

   Or have established, clinically significant coronary and other atherosclerotic vascular disease (meaning at high risk for surgical intervention or for MI, TIA, stroke, if left untreated), including:
   * Angina (stable or unstable)
   * Peripheral arterial disease
   * Atherosclerotic aortic disease
   * Carotid artery disease Or have had
   * CABG (coronary artery bypass graft)
   * PCI (percutaneous coronary intervention with or without stent)
   * Carotid endarterectomy
3. A. If female, subjects are eligible if they are of

   1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
   2. childbearing potential, have a negative pregnancy test at screening, and at least one of the following applies or is agreed to by the subject:

      * Female sterilization or sterilization of male partner
      * Hormonal contraception by oral route, implant, injectable, vaginal ring
      * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year
      * Double barrier method (2 physical barriers or 1 physical barrier plus spermicide)
      * Any other method with published data showing that the lowest expected failure rate is less than 1% per year 4. Able to understand and comply with study procedures required and able and willing to provide written informed consent prior to any study procedures being performed

Exclusion criteria:

1. Any current gastric, esophageal or duodenal ulcer
2. Positive test result for H. pylori at screening 3A. Have had a revascularization procedure (i.e., Coronary Artery Bypass Graft, Percutaneous Transluminal Coronary Angioplasty, or carotid endarterectomy) less than six months prior to screening

4. Unstable hypertension as judged by the Investigator 5. Uncontrolled diabetes mellitus as judged by the Investigator 6. Unstable cardio- or cerebrovascular disease such that it would endanger the subject if they participated in the trial 7. Clinically significant valvular disease 8. Congestive heart failure or other cardiovascular symptoms according to New York Heart Association (NYHA) Functional Classification III-IV (Appendix 3) 9. History of hypersensitivity to omeprazole or to another proton pump inhibitor 10. History of allergic reaction or intolerance to aspirin and/or a history of aspirin-induced symptoms of asthma, rhinitis, and/or nasal polyps 11. History of serious UGI event, such as bleeding, perforation, or obstruction 12. Gastrointestinal disorder or surgery leading to impaired drug absorption 13. Presence of chronic or uncontrolled acute medical illness, e.g. gastrointestinal disorder (esophageal stricture, severe esophagitis, long-segment Barrett's esophagus, signs and symptoms of gastric outlet obstruction), thyroid disorder and/or infection that would endanger a subject if they were to participate in the study 14. Schizophrenia, uncontrolled bipolar disorder, or severe depression 15. History of alcoholism or drug addiction within a year prior to enrollment in the study 16. Severe hepatic dysfunction (i.e. cirrhosis or portal hypertension) 17. Blood coagulation disorder, including use of systemic anticoagulants such as warfarin or other vitamin K antagonists 18. Any condition that, in the opinion of the Investigator, may either put the subject at risk or influence the results of the study 19. Use of any excluded concomitant medication (see Section 9.2) 20. Screening laboratory ALT or AST value > two times the upper limit of normal 21A. History of renal insufficiency 22. Other than noted specifically, any screening laboratory value that is clinically significant in the Investigator's opinion and would endanger a subject if the subject was to participate in the study 23. Use of an investigational treatment in the 4 weeks before screening 24. History of malignancy, treated or untreated, within the past five years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin 25. Previous participation in another PA32540 clinical research study 26. Subjects, who are employees of the research facility, immediately related to the Investigator, or are in some way under the supervision of the Investigator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pozen, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Goldstein JL, Whellan DJ, Scheiman JM, Cryer BL, Eisen GM, Lanas A, Fort JG. Long-Term Safety of a Coordinated Delivery Tablet of Enteric-Coated Aspirin 325 mg and Immediate-Release Omeprazole 40 mg for Secondary Cardiovascular Disease Prevention in Patients at GI Risk. Cardiovasc Ther. 2016 Apr;34(2):59-66. doi: 10.1111/1755-5922.12172. PMID 26725920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center US study in which 44 sites recruited subjects between November 2009 and May 2010
Pre-assignment Details: Screening for eligibility and wash-out of restricted medications
Groups:
- PA32540 Tablet: 325 mg enteric coated (EC) ASA and 40 mg omeprazole to be taken by mouth once daily
  PA32540: PA32540 tablets contain 325 mg enteric coated (EC) aspirin and 40 mg immediate-release omeprazole to be taken by mouth once daily (QD)
Period: Overall Study
Arm/Group | PA32540 Tablet
Started | 380
Treated | 379
Completed | 292
Not Completed | 88
Not completed — Adverse Event | 51
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 2
Not completed — Misc | 28

BASELINE CHARACTERISTICS:
Population: Overall safety population: the overall safety population consisted of all enrolled subjects who received at least one dose of study drug.
Arm/Group | PA32540 Tablet
Number analyzed (Participants) | 379
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 130
  >=65 years | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 266

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Monitored for Long-term Safety of PA32540
Description: Incidence of adverse events and monitoring vital signs and clinical laboratory values. All AEs were coded into preferred terms according to MedDRA (Medical Dictionary for Regulatory Activities) and classified by system organ class (SOC).
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PA32540 Tablet
Number analyzed (Participants) | 379
participants | 379

2. Secondary Outcome: Most Frequent Treatment Emergent Adverse Events Leading to Study Drug Discontinuation
Description: Most Frequent (≥ 1%) Treatment Emergent Adverse Events by System Organ Class leading to Discontinuation
Time Frame: 12 months
Population: Overall Safety Population. Events were collected by systematic assessment. One subject reported two adverse events leading to discontinuation from the study. SOC from vocabulary, MedDRA (12.1).
Measure: Number; unit: participants
Units Other Than Participants: Number of AEs Leading to Discontinuation
Arm/Group | PA32540 Tablet
Number analyzed (Participants) | 379
Number analyzed (Number of AEs Leading to Discontinuation) | 52
participants
  Subjects with any AE Leading to Discontinuation | 51
  Gastrointestinal disorders | 15
  Neoplasms benign, malignant and unspecified | 7
  Cardiac Disorders | 6
  Investigations | 6

ADVERSE EVENTS:
Time Frame: Informed consent through 12 months plus 28 days for Serious Adverse Events and Randomization through 12 months for all non-serious adverse events.
Arm/Group | PA32540 Tablet
Serious Adverse Events (participants affected / at risk) | 55/379
Other Adverse Events (participants affected / at risk) | 280/379
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA32540 Tablet (N=379)
Angina pectoris (Cardiac disorders) | 4 (5)
Angina unstable (Cardiac disorders) | 3 (3)
Coronary artery disease (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (3)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Melaena (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Subdural haematoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thalmic infarction (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA32540 Tablet (N=379)
Bronchitis (Infections and infestations) | 16 (17)
Upper respiratory tract infection (Infections and infestations) | 16 (19)
Nasopharyngitis (Infections and infestations) | 15 (18)
Sinusitis (Infections and infestations) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 20 (24)
Dyspepsia (Gastrointestinal disorders) | 16 (16)
Nausea (Gastrointestinal disorders) | 16 (20)
Constipation (Gastrointestinal disorders) | 11 (11)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Angina pectoris (Cardiac disorders) | 9 (12)
Dizziness (Nervous system disorders) | 11 (11)
Headache (Nervous system disorders) | 11 (12)
Fatigue (General disorders) | 10 (10)
Oedema peripheral (General disorders) | 10 (11)
Haemoglobin decreased (Investigations) | 9 (9)
Hypertension (Vascular disorders) | 11 (11)
Anaemia (Blood and lymphatic system disorders) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: PI agrees that the first publication will be a multi-center publication of the study results. Following this multi-center publication, PI can publish, present or use any non-confidential study results following Sponsor review and comment.